CLINICAL TRIAL: NCT06394414
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Combination with Serplulimab with or Without Platinum-based Chemotherapy in Selected Subjects with Advanced Solid Tumors
Brief Title: A Phase 1 Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-102-02
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose escalation (Experimental): YL201 in Combination with Serplulimab with or without Platinum-based Chemotherapy
  Interventions: Drug: YL201
- Part2: Cohort Expansion (Experimental): YL201 in Combination with Serplulimab with or without Platinum-based Chemotherapy
  Interventions: Drug: YL201

INTERVENTIONS:
Drug: YL201 — YL201 (High dose, medium dose and low dose; Q3W) in Combination with Serplulimab (4.5mg/kg; Q3W) with or without Platinum(70 mg/m2; Q3W)-based Chemotherapy.
  Other Names: Serplulimab; Platinum

SUMMARY:
This is a phase 1, multicenter, open-label stydy to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Combination with Serplulimab with or without Platinum-based Chemotherapy in Selected Subjects with Advanced Solid Tumors conducted in China. The study will include 2 parts: a dose escalation part (Part 1) followed by a cohort expansion part (Part 2).

Part 1 will estimate the safety, tolerability and MTD/RED(s) of YL201 in combination with serplulimab with or without platinum-based chemotherapy in selected subjects with advanced solid tumors.

Part 2 will estimate the efficacy of YL201 in combination with serplulimab with or without platinum-based chemotherapy in selected subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1) Informed of the study before the start of the study and voluntarily sign their name and date on the informed consent form (ICF).

  2) Subjects will be enrolled in the dose-escalation phase: Advanced solid tumors, like NPC, SCLC and etc.

  3) Subjects will be enrolled in the dose-expansion phase: NPC, SCLC, NSCLC and other advanced cancer.

  4) According to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, there must be at least one extracranial measurable lesion.

  5) Archived or fresh tumor tissue samples can be provided. 6) Within 7 days before the first dose, organ and bone marrow functions must meet the requirements.

  7) Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1 by the United States of America standards.

  8) Female subjects of childbearing potential must agree to use highly effective contraception measures from screening throughout the duration of the study and for at least 6 months after the last dose of the study drug. Male subjects must agree to use highly effective contraception measures from screening throughout the duration of the study and for at least 6 months after the last dose of the study drug.

  9) Subjects with expected survival ≥ 3 months. 10) Capable and willing to comply with the study protocol's scheduled visits and procedures.

Exclusion Criteria:

* 1) Suitable for local radical treatment. 2) Previous Drug therapy targeting B7H3. 3) Previous Drug therapy with topoisomerase I inhibitors or ADCs composed of topoisomerase I inhibitors.

  4) Prior treatment with anti-PD-(L)1, other immune checkpoint inhibitors, immune checkpoint agonists, or immunocellular therapies and other therapies targeting tumor immunity mechanisms.

  5) Toxicity from previous anticancer treatments has not resolved. 6) Concurrent enrollment in another clinical study. 7) Inadequate washout period for prior anticancer treatment before the first dose of study drug.

  8) Underwent major surgery (excluding diagnostic surgery) or suffered serious trauma.

  9) Received allogeneic stem cell or solid organ transplant. 10) Active autoimmune diseases requiring systemic treatment. 11) Received systemic steroids. 12) Metastases to meninges or carcinomatous meningitis. 13) Brain metastasis or spinal cord compression. 14) Uncontrolled or clinically significant cardiovascular disease. 15) Clinically significant concomitant pulmonary disease. 16) With uncontrolled third-space fluid. 17) History of gastrointestinal perforation and / or fistula within 6 months prior to the first dose.

  18) Serious Infection prior to the first dose. 19) Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

  20) Any other primary malignancy before the first dose of study drug. 21) A history of severe hypersensitivity reactions to the investigational product, inactive ingredients in the formulation, or other monoclonal antibodies.

  22) Women who are breastfeeding or pregnant as confirmed by pregnancy tests performed within 3 days before the first dose.

  23) Any illness, medical condition, organ system dysfunction, or social situation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2030-04-29 (Estimated)

PRIMARY OUTCOMES:
Evaluate the AEs in YL201 combination with serplulimab with or without platinum-based chemotherapy in advanced solid tumors | Approximately within 36 months
  AE: Adverse Event
To determine the MTD/RED of YL201 in combination with serplulimab with or without platinum-based chemotherapy in advanced solid tumors | Approximately within 36 months
  maximum tolerated dose (MTD), recommended expansion dose (RED)
To evaluate the efficacy of YL201 in combination with serplulimab with or without platinum-based chemotherapy in advanced solid tumors based on ORR | Approximately within 36 months
  objective response rate (ORR)
To determine the RP2D of YL201 in combination with serplulimab with or without platinum-based chemotherapy in advanced solid tumors based on ORR | Approximately within 36 months
  recommended Phase 2 dose (RP2D)

SECONDARY OUTCOMES:
To evaluate the AUC of YL201 combination therapy | Approximately within 36 months
  area under the curve (AUC)
To evaluate the Cmax of YL201 combination therapy | Approximately within 36 months
  peak concentration (Cmax)
To evaluate the Ctrough of YL201 combination therapy | Approximately within 36 months
  trough concentration (Ctrough)
To evaluate the CL of YL201 combination therapy | Approximately within 36 months
  clearance rate (CL)
To evaluate the Vd of YL201 combination therapy | Approximately within 36 months
  volume of distribution (Vd)
To evaluate the t1/2 of YL201 combination therapy | Approximately within 36 months
  half-life time (t1/2)
To evaluate the DpR of YL201 combination therapy | Approximately within 36 months
  depth of response (DpR); assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
To evaluate the DCR of YL201 combination therapy | Approximately within 36 months
  disease control rate (DCR); assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
To evaluate the DoR of YL201 combination therapy | Approximately within 36 months
  duration of response (DoR); assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
To evaluate the TTR of YL201 combination therapy | Approximately within 36 months
  time to response (TTR); assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
To evaluate the PFS of YL201 combination therapy | Approximately within 36 months
  progression-free survival (PFS); assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
To evaluate the OS of YL201 combination therapy | Approximately within 36 months
  Overall survival (OS)
To evaluate the immunogenicity of YL201 combination therapy | Approximately within 36 months
  Incidence of anti-YL201 antibodies
To assess the expression level of B7H3 and PD-L1 in Tumor tissue | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijinig
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Provincial Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College HuaZhong University of Science Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changhua, Jilin
  - Liaoning Provincial Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Linyi Central Hospital, Linyi, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Sichuan, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No